CLINICAL TRIAL: NCT00176423
Title: Adjunctive Galantamine for Treatment of Cognitive Impairments in Patients With Schizophrenia
Brief Title: Efficacy Study of Galantamine for Cognitive Impairments in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Stanley Medical Research Institute (Other); Ortho-McNeil Neurologics, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Buchanan, Director, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01T-411
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; acetylcholine; cognitive impairments; attention; processing speed; sensory gating; eye-tracking
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- galantamine (Experimental): galantamine, 24mgs, p.o., qday
  Interventions: Drug: galantamine
- placebo (Placebo Comparator): placebo, 3 tablets, p.o., qday
  Interventions: Drug: galantamine

INTERVENTIONS:
Drug: galantamine — see arm/group description

SUMMARY:
The purpose of this study is to examine whether adjunctive galantamine is effective in the treatment of cognitive impairments in patients with schizophrenia.

DETAILED DESCRIPTION:
Patients with schizophrenia are characterized by a broad range of neurocognitive abnormalities. These include impairments in attention; eye-tracking; visual and verbal memory; working memory; processing speed; and sensory gating, as measured by P50. These impairments are major determinants of poor functional outcome in patients with schizophrenia. Conventional antipsychotics have limited effects on these impairments. Second generation antipsychotics (SGAs) may have modest benefits for cognitive function, but whether this represents a direct cognitive enhancing effect has not been established. Regardless, patients continue to exhibit pronounced cognitive impairments despite adequate new generation antipsychotic treatment. Adjunctive pharmacotherapy may offer a viable approach for the treatment of cognitive impairments. Adjunctive agents can be used to modulate specific neurotransmitter systems that are hypothesized to be involved in the pharmacology of cognitive functions.

Acetylcholine acts at muscarinic and nicotinic cholinergic receptors. These receptors are broadly distributed through the brain, including the neocortex, hippocampus, and basal ganglia. Cholinergic mechanisms have been implicated in the regulation of attention, memory, processing speed, and sensory gating processes; processes which are impaired in patients with schizophrenia. Nicotine has previously been shown to improve sensory gating, as measured by P50, and eye-tracking in patients with schizophrenia. The gene for the alpha-7 nicotinic receptor, which is hypothesized to be the nicotinic receptor involved in sensory gating regulation, has also been shown to be linked to schizophrenia.

Galantamine (Trade name: Reminyl) is a new FDA-approved selective acetylcholinesterase inhibitor (AChEI), which may also allosterically modulate nicotinic receptors, enhance receptor sensitivity, and increase nicotinic receptor density. Galantamine is marketed by Janssen Research Foundation. In animal models of aging, galantamine enhanced long-term potentiation, ameliorated learning impairments, and elevated the number of nicotinic receptors in the hippocampus and neocortex. In placebo-controlled studies, galantamine has been shown to not only delay deterioration but to improve cognitive function in patients with Alzheimer's disease. There is also preliminary evidence that galantamine may ameliorate positive psychotic symptoms in these patients.

AChEIs have not been extensively studied in patients with schizophrenia. We have conducted a 6-week open-labeled pilot study of adjunctive donepezil in patients treated with olanzapine for a minimum of 6 months. Fifteen patients entered the study and 14 patients completed the study. One patient withdrew with a complaint of sedation. The demographic characteristics of the patients who completed the study were: mean (SD) age: 43.1 6.6; 71% male; 78% caucasian; and mean (SD) duration of illness: 24.7 7.2. The mean (SD) olanzapine dose was 25.7 11.9 mg/day. Two patients were receiving benzodiazepines, two were receiving antidepressants, and one was receiving valproic acid. Donepezil resulted in a modest improvement in sensory gating. Nine patients had abnormal P50 at baseline, which normalized for five patients following treatment. Donepezil had a more pronounced effect on neuropsychological test performance, with large and significant effect sizes observed for the visual memory (effect size (ES)=.57) and manual dexterity (ES=.93) measures. There were moderate improvements on the verbal recall memory (ES=0.46) and processing speed (ES=0.48) measures. The only cognitive measure that did not change with treatment was a measure of attention. There were no significant changes in either positive symptom (mean (SD), baseline: 9.3 3.8; week 6: 8.2 3.8; t=-1.55, df=14, p=.14) or negative symptom (mean(SD), baseline: 29.7 10.9; week 6: 30.0 12.6; t=0.15, df=14, p=.88) measures.

The results of this study suggest that adjunctive AChEIs may be an effective treatment for cognitive impairments in patients with schizophrenia. Moderate to large effect size improvements were observed on verbal and visual memory, processing speed, and manual dexterity measures. Patients exhibited a greater than 20% increase in suppression of their P50 response to repeated auditory stimuli. There was no effect of donepezil on a measure of attention. Donepezil was well tolerated; only one patient dropped out of the study and nine of the remaining subjects chose to continue on the drug beyond the protocol. An important aspect of the study was that cognitive function improvement occurred in the context of concurrent olanzapine treatment, which is reported to improve P50 and cognitive function (Purdon et al, 2000; Light et al, 2000). Thus, donepezil was able to further enhance cognitive function in patients who may have already benefitted from olanzapine treatment.

The primary study objectives are:

1. To examine whether adjunctive galantamine is more effective than placebo for neuropsychological measures of attention, verbal and visual memory, working memory, processing speed, and manual dexterity.
2. To examine whether adjunctive galantamine is more effective than placebo for evoked potential measures of sensory gating (i.e., P50) and attention (i.e., P300 and Gamma Band Response (GBR)) and smooth pursuit eye movement.

We hypothesize that galantamine will have a significant benefit for these cognitive behaviors based on the role of acetylcholine in the regulation of these behaviors; our pilot study with donepezil which demonstrated that AChEIs may have a beneficial effect for verbal and visual memory, processing speed, and manual dexterity; and previous studies that have shown acute nicotine administration to normalize P50 and eye-tracking in patients with schizophrenia.

The secondary study objectives are:

1. To examine whether adjunctive galantamine is more effective than placebo for positive symptoms and negative symptom measures.
2. To examine whether adjunctive galantamine is more likely than placebo to cause nausea, vomiting, diarrhea, anorexia, weight loss, or dizziness, i.e., common side effects associated with AChEI treatment.
3. To examine whether galantamine is more likely than placebo to cause an increase in either extrapyramidal symptoms or dyskinetic movements.
4. To examine whether galantamine is more effective than placebo for reducing smoking behavior.

We hypothesize that there will not be a significant difference between galantamine and placebo for positive and negative symptoms based on our donepezil pilot study. We hypothesize that galantamine will be associated with an increased incidence of AChEI associated side effects. We hypothesize that there will not be a significant difference between galantamine and placebo for either extrapyramidal symptoms or dyskinetic movements.

Study Design and Methods: The proposed study is a randomized, parallel group, double-blind comparison of adjunctive galantamine or placebo. The sample will consist of 90 clinically stable inpatients and outpatients with DSM-IV schizophrenia or schizoaffective disorder. There will be a 2-week stabilization phase, a 12-week treatment phase, and an optional 6-month open-label phase. In the 2-week stabilization phase, patients will undergo baseline symptom, medical, safety, antipsychotic level, and neurocognitive assessments. In the 12-week treatment phase, patients will be randomized to either galantamine or placebo. Patients will receive biweekly symptom, side effect, and vital sign assessments. At the end of study (12 weeks), laboratory tests, EKG, antipsychotic levels, and neurocognitive assessments will be repeated. Patients will be monitored at the 3-month and 6-month points of the open-labeled phase, during which they will receive laboratory tests, EKG, and side effect review. At the end of the 6-month open-labeled phase, patients will again be asked to participate in symptom ratings and neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV diagnosis of either schizophrenia or schizoaffective disorder.
2. Males and females
3. Age: 18 and 60
4. Caucasian or Non-Caucasian
5. Subjects will be currently treated with one of the following new generation antipsychotics: olanzapine, risperidone, quetiapine, ziprasidone, or aripiprazole.
6. Subjects will meet a priori criteria for cognitive impairment severity. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) will be used to determine the level of cognitive impairment. Patients will meet entry criteria if they have a RBANS total score of 90 or less (one standard deviation below the normal control mean).

Exclusion Criteria:

1. History of an organic brain disease
2. History of DSM-IV alcohol or substance abuse (within the last month), or DSM-IV alcohol or substance dependence (within the last six months).
3. Pregnant women and women taking oral contraceptives (because of the theoretical risk of breakthrough ovulation).
4. Current treatment with galantamine or other acetylcholinesterase inhibitor (e.g. donepezil)
5. History of a second or third degree atrioventricular (AV) block.
6. Persons with chronic medical conditions, which are unstable.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, M.D., Principal Investigator — University of Maryland Baltimore School of Medicine, Maryland Psychiatric Research Center
Locations (1):
- Maryland Psychiatric Research Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Buchanan RW, Conley RR, Dickinson D, Ball MP, Feldman S, Gold JM, McMahon RP. Galantamine for the treatment of cognitive impairments in people with schizophrenia. Am J Psychiatry. 2008 Jan;165(1):82-9. doi: 10.1176/appi.ajp.2007.07050724. Epub 2007 Nov 6. PMID 17986678

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of people who signed informed consent was "117". Thirty-one participants who signed informed consent did not complete the Evaluation Phase of the study and were not randomized. Eight-six (86) participants completed the Evaluation Phase of the study and were randomized.
Period: Overall Study
Arm/Group | Galantamine | Placebo
Started | 42 | 44
Completed | 35 | 38
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine | Placebo | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 44 | 86
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 37 | 37 | 74
Region of Enrollment [Number; unit: participants]
  United States | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Overall Cognitive Improvement Z-score
Description: Participants were administered an eight-test neuropsychological test battery at baseline and end-of-study. The battery included the following tests: working memory: WAIS-III Letter-Number Sequencing and Brief Assessment of Cognition in Schizophrenia Number Sequencing; verbal memory: California Verbal Learning Test (CVLT); visual memory: Brief Visuospatial Memory Test (BVMT); motor speed: Grooved Pegboard; processing speed: WAIS-III Digit Symbol and WAIS-III Symbol Search; and the Gordon Diagnostic System CPT. Alternate forms of the CVLT and BVMT were used for the two test occasions. For each neuropsychological test, participant scores were converted to z-scores: z = (score - baseline mean)/baseline SD. For the primary outcome measure, an overall composite z-score was computed from the average of the individual test z-scores. A positive z-score would reflect better performance compared to baseline; a negative z-score would reflect worse performance compared to baseline.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 35 | 38
z-score
  Week 0 | 0.03 (0.64) | -0.03 (0.05)
  Week 12 | 0.15 (0.68) | 0.61 (0.55)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: ECG Changes From Baseline to 12 Weeks.
Description: Three measures were examined: PR interval, QRS interval, and QTc interval. The three measures were derived from a standard 12-lead ECG recording.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 42 | 44
msec
  PR interval | 25.7 (56.0) | 3.0 (12.0)
  QRS interval | 11.4 (25.1) | -1.6 (11.7)
  QTc interval | 3.03 (28.89) | 3.03 (27.68)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

3. Secondary Outcome: Simpson Angus Scale (SAS) Total Score
Description: The SAS total were calculated by adding scores from scales #1-#11. Each scale ranges from "0=None/Normal" to "4=Extreme/Severe". The minimum total score is 0 and the maximum score is 44. Higher scores indicate a more severe extrapyramidal side effect rating.
Time Frame: 12 weeks (Week 12 - Week 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Week 0 | 1.4 (1.8) | 1.6 (2.1)
  Week 12 | 1.1 (1.8) | 1.6 (1.9)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

4. Secondary Outcome: Abnormal Involuntary Movement Scale (AIMS)
Description: Change in AIMS Total Score: Frequencies of Maximum Within-Participant Increases (worsening) from Baseline by Treatment Group. Total score calculated by adding scores from scales #1-#10. Each scale ranges from "0=None" to "4=Severe". The minimum total AIMS score is 0 and the maximum score is 40. Higher scores indicate a more severe abnormal involuntary movement rating.
Time Frame: 12 weeks (Week 12 - Week 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 42 | 44
score on a scale
  Week 0 | 2.0 (3.1) | 2.1 (3.1)
  Week 12 | 2.1 (3.0) | 1.6 (3.0)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Galantamine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/44
Other Adverse Events (participants affected / at risk) | 2/42 | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine (N=42) | Placebo (N=44)
hospitalization due to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine (N=42) | Placebo (N=44)
worsening of psychiatric symptoms (Psychiatric disorders) | 1 | 1
increased alcohol consumption (Social circumstances) | 1 | 0
dizziness (Ear and labyrinth disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes